CLINICAL TRIAL: NCT03236935
Title: Phase Ib Trial of L-NMMA in Combination with Pembrolizumab in Patients with Melanoma, Non-Small Cell Lung Cancer, Head and Neck Squamous Cell Carcinoma, Classical Hodgkin Lymphoma, Urothelial Carcinoma, Cervical Cancer, Esophageal Cancer, Gastric Cancer, Hepatocellular Carcinoma, Merkel Cell Carcinoma, Primary Mediastinal Large B-cell Lymphoma, Renal Cell Carcinoma, Small Cell Lung Cancer, Microsatellite Instability-High/Mismatch Repair Deficient Cancer, or for the Treatment of Adult Patients with Unresectable or Metastatic Tumor Mutational Burden-High Solid Tumors
Brief Title: Phase Ib of L-NMMA and Pembrolizumab
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Jun Zhang, Principal Investigator, The Methodist Hospital Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00017492
Record Dates: First submitted 2017-07-28; First posted 2017-08-02 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2024-08

CONDITIONS: Non-Small Cell Lung Cancer; Malignant Melanoma; Head and Neck Squamous Cell Carcinoma; Classical Hodgkin Lymphoma; Urothelial Carcinoma Bladder; DNA Repair-Deficiency Disorders
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Melanoma; Squamous Cell Carcinoma of Head and Neck; DNA Repair-Deficiency Disorders | interventions — omega-N-Methylarginine; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- L-NMMA Plus Pembrolizumab (Experimental): L-NMMA and pembrolizumab will be administered for 6 cycles. Cycle length will be 21 days. L-NMMA will be administered as a 2-hour intravenous (IV) infusion on Days 1-5 at each cycle. The dose levels of L-NMMA are as follows: Dose Level -1, 12.5 mg/kg; Dose Level 0 (starting dose), 15.0 mg/kg; and Dose Level 1, 20 mg/kg. L-NMMA dose will escalate/de-escalate based on the occurrence of dose-limiting toxicities. Pembrolizumab at a fixed dose of 200 mg will be IV infused over 30 minutes on Day 5 at each cycle. Pembrolizumab will be administered 1 hour after L-NMMA infusion on Day 5 at each cycle. Subjects without disease progression after 6 cycles of L-NMMA and pembrolizumab will continue pembrolizumab until disease progression or unacceptable AEs.
  Interventions: Drug: L-NMMA; Drug: Pembrolizumab

INTERVENTIONS:
Drug: L-NMMA — pan-nitric oxide synthase inhibitor
  Other Names: NG-monomethyl-L-arginine
Drug: Pembrolizumab — PD-1 inhibitor
  Other Names: Keytruda

SUMMARY:
The purpose of this Phase Ib study is to test the safety of NG-monomethyl-L-arginine (L-NMMA) and pembrolizumab when used together in participants with melanoma, non-small cell lung cancer (NSCLC), head and neck squamous cell carcinoma (HNSCC), classical Hodgkin lymphoma (cHL), urothelial carcinoma, Cervical Cancer, Esophageal Cancer, Gastric Cancer, Hepatocellular Carcinoma, Merkel Cell Carcinoma, Primary Mediastinal Large B-cell Lymphoma, Renal Cell Carcinoma, Small Cell Lung Cancer, microsatellite instability-high (MSI-H)/mismatch repair deficient (dMMR) cancer or for the Treatment of Adult Patients with Unresectable or Metastatic Tumor Mutational Burden-High Solid Tumors. Pembrolizumab is a type of treatment that stimulates the immune system to attack cancer cells. The immune system is normally the body's first defense against threats like cancer. However, sometimes cancer cells produce signals like programmed death-1 (PD-1) that prevent the immune system from detecting and killing them. Pembrolizumab blocks PD-1 so your immune system can detect and attack cancer cells. To help further boost the cancer-fighting ability of your immune system, L-NMMA will be used along with pembrolizumab. L-NMMA is a nitric oxide synthase inhibitor. The presence of nitric oxide synthase in the area around the cancer cells blocks the cancer-fighting ability of the immune system. Thus, the use of L-NMMA and pembrolizumab together may make the immune system work harder to attack and destroy the cancer cells.

DETAILED DESCRIPTION:
The purpose of this Phase Ib study is to test the safety of NG-monomethyl-L-arginine (L-NMMA) and pembrolizumab when used together in participants with melanoma, non-small cell lung cancer (NSCLC), head and neck squamous cell carcinoma (HNSCC), classical Hodgkin lymphoma (cHL), urothelial carcinoma, Cervical Cancer, Esophageal Cancer, Gastric Cancer, Hepatocellular Carcinoma, Merkel Cell Carcinoma, Primary Mediastinal Large B-cell Lymphoma, Renal Cell Carcinoma, Small Cell Lung Cancer, microsatellite instability-high (MSI-H)/mismatch repair deficient (dMMR) cancer or for the Treatment of Adult Patients with Unresectable or Metastatic Tumor Mutational Burden-High Solid Tumors. Pembrolizumab is a type of treatment that stimulates the immune system to attack cancer cells. The immune system is normally the body's first defense against threats like cancer. However, sometimes cancer cells produce signals like PD-L1 that prevent the immune system from detecting and killing them. Pembrolizumab blocks programmed death-1 (PD-1) so your immune system can detect and attack cancer cells. To help further boost the cancer-fighting ability of your immune system, L-NMMA will be used along with pembrolizumab. L-NMMA is a nitric oxide synthase inhibitor. The presence of nitric oxide synthase in the area around the cancer cells blocks the cancer-fighting ability of the immune system. Thus, the use of L-NMMA and pembrolizumab together may make the immune system work harder to attack and destroy the cancer cells.

In this study, up to 3 different doses of L-NMMA will be studied (12.5, 15, and 20 mg/kg). Participants will only receive one of the three L-NMMA doses. The first several study participants will receive the 15 mg/kg dose. If the 15 mg/kg dose of L-NMMA causes serious side effects, L-NMMA will be given to other study participants at the lower dose of 12.5 mg/kg. If the 15 mg/kg dose of L-NMMA does not cause serious side effects, L-NMMA will be given to other study participants at the higher dose of 20 mg/kg. All study participants will be given the same dose of pembrolizumab (200 mg). This study will allow us to see the highest dose of L-NMMA that can be used safely with pembrolizumab in participants with melanoma, NSCLC, HNSCC, cHL, urothelial carcinoma, or MSI-H/dMMR cancer.

ELIGIBILITY:
Inclusion Criteria:

* Female or male aged ≥ 18 years on the day of informed consent signing;
* Has histologically confirmed metastatic melanoma that is treatment naïve or has relapsed after or is refractory to ipilimumab or BRAF inhibitor (if BRAF mutation-positive), OR histologically confirmed metastatic NSCLC that has high programmed death-ligand 1 (PD-L1) expression (tumor proportion score [TPS] ≥50%) with no epidermal growth factor receptor (EGFR) or anaplastic lymphoma kinase (ALK) genomic tumor aberrations or histologically confirmed metastatic NSCLC that is PD-L1 positive (TPS ≥1%) and has progressed on or after platinum-containing therapy (subjects with NSCLC harboring EGFR/ALK genomic aberrations must have received an FDA-approved targeted therapy for these aberrations) OR histologically confirmed HNSCC that has relapsed after or is refractory to platinum-containing chemotherapy, OR histologically confirmed cHL that has relapsed after three or more lines of therapy or is refractory to treatment OR histologically confirmed locally advanced or metastatic urothelial carcinoma that is not eligible for platinum-containing chemotherapy or that has relapsed after or is refractory to platinum-containing chemotherapy OR histologically confirmed advanced, PD-L1-positive cervical cancer with disease progression on or after chemotherapy that is not eligible for platinum-containing chemotherapy or that has relapsed after or is refractory to platinum-containing chemotherapy OR histologically confirmed recurrent, locally advanced, or metastatic, squamous cell carcinoma of the esophagus (ESCC) whose tumors express PD-L1 (Combined Positive Score [CPS] ≥10), as determined by an FDA-approved test, with disease progression after one or more prior lines of systemic therapy.

OR histologically confirmed recurrent, locally advanced, or metastatic Gastric Cancer, with disease progression on or after two or more systemic therapies, including fluoropyrimidine- and platinum-containing chemotherapy and, if appropriate, HER2/neu-targeted therapy, and whose tumors express programmed death-ligand 1 (PD-L1), as determined by an FDA-approved test.

OR histologically confirmed hepatocellular carcinoma (HCC) who have been previously treated with sorafenib. recurrent locally advanced or metastatic MCC who had not received prior systemic therapy for their advanced disease OR histologically confirmed recurrent, locally advanced or metastatic Merkel Cell Carcinoma (MCC) who had not received prior systemic therapy for their advanced disease OR histologically confirmed advanced renal cell carcinoma (RCC) first-line treatment.

OR histologically confirmed metastatic small cell lung cancer (SCLC) with disease progression on or after platinum-based chemotherapy and at least one other prior line of therapy.

OR histologically confirmed refractory primary mediastinal large B-cell lymphoma (PMBCL), who have relapsed after two or more prior lines of therapy.

OR MSI-H or dMMR unresectable or metastatic cancer that has relapsed after prior treatment and has no satisfactory alternative treatment options.

OR adult patients with unresectable or metastatic tumor mutational burden-high (TMB-H) [≥10 mutations/megabase (mut/Mb)] solid tumors;

* Measurable disease based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1;
* Eastern Cooperative Oncology Group performance status of 0-2;
* Life expectancy ≥ 6 months;
* Adequate organ function:

Absolute neutrophil count ≥1,500/mm3, platelets ≥100,000/mm3, hemoglobin ≥9 g/dL (transfusion permitted), serum creatinine OR measured or calculated creatinine clearance ≤1.5 X upper limit of normal (ULN) OR ≥60 mL/min for subject with creatinine levels > 1.5 X institutional ULN, serum total bilirubin ≤ 1.5 X ULN OR direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN, alanine transaminase and aspartate transaminase ≤ 2.5 X ULN OR ≤ 5 X ULN for subjects with liver metastases, albumin >2.5 mg/dL, International normalized ratio or prothrombin time ≤1.5 X ULN, and activated partial thromboplastin time ≤1.5 X ULN;

* Cardiac ejection fraction of ≥ 45%;
* Female subjects of childbearing potential should have a negative serum pregnancy (beta-human chorionic gonadotropin) within 7 days prior to receiving the first dose of trial treatment and should not be lactating;
* Female subjects of childbearing potential must be willing to use an adequate method of contraception for the course of the trial through 120 days after the last dose of trial treatment;
* Male subjects of childbearing potential must be willing to use an adequate method of contraception for the course of the trial through 120 days after the last dose of trial treatment;
* Willing and able to provide written informed consent/assent for the trial.

Exclusion Criteria:

* History of poorly controlled hypertension (defined as systolic blood pressure >150 mmHg);
* History of New York Heart Association class III or greater cardiac disease;
* History of myocardial infarction, stroke, ventricular arrhythmia, or symptomatic conduction abnormality within the past 12 months;
* History of congenital QT prolongation;
* Absolute corrected QT interval of >480 milliseconds in the presence of potassium >4.0 milliequivalent/L and magnesium >1.8 mg/dL;
* Currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of the trial treatment;
* Concurrent use of medications that interact with nitrate/nitrites;
* Concurrent use of any complementary or alternative medicines;
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment;
* Known history of active tuberculosis (Bacillus Tuberculosis);
* Hypersensitivity to L-NMMA, pembrolizumab, or any of their excipients;
* Has had a prior anticancer monoclonal antibody within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier;
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent;
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
* Has known active central nervous system metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least 4 weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability;
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease-modifying agents, corticosteroids or immunosuppressive drugs);
* History of non-infectious pneumonitis that required steroids or current pneumonitis;
* Has an active infection requiring systemic therapy;
* History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator;
* Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial;
* Is pregnant or breastfeeding, or expecting to conceive a child within the projected duration of the trial, starting with the prescreening or screening visit through 120 days after the last dose of trial treatment;
* Received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent;
* Known history of human immunodeficiency virus;
* Has known active hepatitis B or hepatitis C;
* Received a live vaccine within 30 days of planned start of the trial treatment;
* Unwilling or unable to comply with the trial protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-08-03 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2025-12-28 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | 18 weeks
  Assess the MTD of L-NMMA in combination with pembrolizumab

SECONDARY OUTCOMES:
Dose-limiting toxicities (DLTs) and other adverse events | 18 weeks
  Describe the DLTs and other adverse events associated with the combination of L-NMMA and pembrolizumab, as assessed by the Common Terminology Criteria for Adverse Events V4.03
Recommended Phase 2 dose (RP2D) of L-NMMA in combination with pembrolizumab | 18 weeks
  Determine the RP2D of L-NMMA in combination with pembrolizumab based on the occurrence of DLTs and MTD determination
Antitumor activity | 18 weeks
  Assess the antitumor activity of L-NMMA in combination with pembrolizumab, as assessed by the RECIST 1.1
Plasma concentrations of L-NMMA when combined with pembrolizumab | 18 weeks
  Measure plasma concentrations of L-NMMA over time

CONTACTS AND LOCATIONS:
Overall Officials: Jun Zhang, M.D., Principal Investigator — Houston Methodist Cancer Center
Locations (1):
- Houston Methodist Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No